CLINICAL TRIAL: NCT03408665
Title: Phase II Study, Stratified, Non-randomized, Estimating SBRT Efficiency and Toxicity in Primary and Secondary Liver Tumors
Brief Title: Stereotactic Body Radiation Therapy (SBRT) Efficiency and Toxicity in Liver Cancer
Acronym: STEREOLIVER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Canceropôle Nord Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STEREOLIVER-1704
Record Dates: First submitted 2018-01-04; First posted 2018-01-24 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Liver Cancer; Liver Metastases
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SBRT (Experimental): Stereotaxic Body Radiation Therapy administred in 3 to 6 fractions.
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — 3 sessions at least, up to 6. Neither specifc device is imposed.

SUMMARY:
Intervention research involving the human person, phase II, prospective, multicentric, non-randomized and multi-cohort study. The eligibility criteria are broad, on purpose, so every patient, able to be treated by SBRT and unable to participate in another trial (non eligible patient or non included centers), can be included in this national study, in a prospective way.

DETAILED DESCRIPTION:
Patients will first go through an inclusion check-up consisting of:

* a clinical exam: disease history, previous treatments, weight, height, patient's performance status (ECOG) and HCC status.
* a biological test: biochemical (total bilirubin, ASAT-ALAT, LDH, albumin, alkaline phosphatases, GGT), hematological (if the patient is going to receive a fiducial), alphafoetoprotein (for HCC) and pregnancy test (if applicable)
* a tumor assessment: using a CT-scan or a MRI and using RECIST or mRECIST (if HCC), plus other morphological exams if judged useful by the investigator This check-up has to be realized within 28 days before inclusion. Then, the use of fiducial is optional.

Before the beginning of the treatment, a pre-therapeutic check-up is done:

* the inclusion check-up has to be done a second time if the treatment begins more than 28 days after the first one
* Tracking scanner.

The SBRT treatment is done in 3 to 6 times and no specific SBRT techniques are asked for, the investigator can choose according to the center habits.

After the treatment, a follow-up will be realized at 3, 6, 9, 12, 18, 24, 30 and 36 months and then once a year until the last patient included reach their 36th month of follow-up. The follow-up check-up consists of a clinical exam, biological test, tumor assessment and tolerance assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* With primary or secondary liver tumor and matching one of the following situations:
* Liver Metastasis (LM): anatomopathologic diagnosis of the primary tumor
* Hepatocellular Carcinoma (HCC): diagnosis achieved through biopsy or through non-invasive methods approved by AASLD criteria (Bruix, 2011)
* Cholangiocarcinoma (CC): diagnosis achieved through biopsy
* Other primitive hepatic tumor achieved through biopsy
* Meet the requirements for SBRT treatment:
* Liver Metastasis (LM): oligometastatic disease
* Hepatocellular Carcinoma (HCC): non eligible lesion to curative surgery
* Cholangiocarcinoma (CC): nodular lesion
* Other primitive hepatic tumor: non eligible lesion to curative surgery
* Able to receive a SBRT treatment according to the multidisciplinary consultation meeting
* Tumor assessable with CT-scan or MRI according to mRECIST in HCC or Recist 1.1 in other situations
* Affiliation to the National Social Security System
* With informed and signed consent

Exclusion Criteria:

* Eligibility to a curative surgery according to the multidisciplinary consultation meeting
* Contraindication to SBRT (especially Cirrhose Child C)
* Pregnant or breastfeeding women
* Patient Under guardianship or tutorship
* Impossibility to submit at the study procedures due to geographic, social or mental reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
SBRT efficiency in term of L-PFS for patient who are to be treated with SBRT in patients with primitive hepatic tumor of hepatic metastatis | From baseline to 36 months following up.
  Local progression-free survival (L-PFS) thanks to Kaplan-Meier method from registration date to date of local progressive disease.

SECONDARY OUTCOMES:
Estimate the SBRT efficiency in a prospective way, in term of local progression-free survival (L-PFS) for patient treated with SBRT in the 4 considered clinical situations. | From baseline to 36 months following up.
  Local progression-free survival (L-PFS) thanks to Kaplan-Meier method from registration date to date of local progressive disease.
Describe the different SBRT techniques used in the study for liver tumor. | From baseline to 36 months following up.
  Description of SBRT techniques used.
Determine the SBRT feasibility by comparison of planned SBRT to performed SBRT. | From baseline to 36 months following up.
  Description of reasons leading to SBRT scheme modification or interruption.
Estimate the SBRT efficiency in a prospective way, in term of overall survival (OS) in the 4 considered clinical situations. | From baseline to 36 months following up.
  Overall survivall thanks to Kaplan-meier method, from registration date to date of death.
Estimate the SBRT efficiency in a prospective way, in term of progression-free survival (PFS) in the 4 considered clinical situations. | From baseline to 36 months following up.
  Progression-free survival (PFS) thanks to Kaplan-Meier method from registration date to date of progressive disease.
Assess the immediate and delayed toxicity. | From baseline to 36 months following up.
  Description of toxicity associated to SBRT or the fiducial use thanks to NCI-CTCAE v4.0.
Estimate the quality-adjusted survival (Q-TWiST) for patients in each of the 4 considered clinical situations. | From baseline to 36 months following up.
  Q-TWIST consists in 3 clinical states: time in toxicity before progressive disease, time in progressive disease, time without toxicity nor progressive disease.
Estimate the proportion of patients for whom an hospitalization is required. | From baseline to 36 months following up.
  during the treatment and until 3 months after and the cumulative duration of the hospitalization over those 3 months.
Estimate the impact of the different SBRT techniques on SBRT efficacy according to L-PFS. | From baseline to 36 months following up.
  Estimation of impact of SBRT technique used on SBRT efficacy according to L-PFS.
Estimate the impact of the different SBRT techniques on SBRT efficacy according to PFS. | From baseline to 36 months following up.
  Estimation of impact of SBRT technique used on SBRT efficacy according to PFS.
Estimate the impact of the different SBRT techniques on SBRT efficacy according to OS. | From baseline to 36 months following up.
  Estimation of impact of SBRT technique used on SBRT efficacy according to OS.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier MIRABEL, MD, Principal Investigator — Centre Oscar Lambret
Locations (7):
- France (7):
  - Centre Oscar Lambret, Lille, Nord
  - Centre Léonard de Vinci, Dechy
  - Institut Régional du Cancer de Montpellier, Montpellier
  - Institut de Cancérologie Paris Nord, Sarcelles
  - Centre Paul Strauss, Strasbourg
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No